CLINICAL TRIAL: NCT05705011
Title: Frailty, Cognitive Function and Health-related Quality of Life in Older Adults With Advanced Chronic Kidney Disease: Mortality and Dialysis Initiation, a Prospective Cohort Study.
Brief Title: Frailty, Cognitive Function and Health-related Quality of Life in Older Adults With Advanced Chronic Kidney Disease.
Status: Completed | Type: Observational
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Hani Hussien, Doctor, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: Nephrogeriatrics
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: CKD Stage 4; CKD Stage 5; Frailty; Cognitive Impairment
Keywords: CKD; FRAILTY; HRQOL
MeSH Terms: conditions — Renal Insufficiency, Chronic; Frailty; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study explores the impact of cognitive impairment and frailty in older adults with advanced chronic kidney disease ].

The main question[s] it aims to answer are:

* What determines the time to initiate dialysis? Cognitive impairment or frailty?
* What does predict the time to death? Presence of frailty or cognitive impairment?
* What does correlate strongly with time-low health-related quality of life? frailty or cognitive impairment?

ELIGIBILITY:
Inclusion Criteria:

* Patients age 65 years or older.
* CKD stage 4 and 5 who were identified by two consecutive measurements of estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 separated by more than 3 months.

Exclusion Criteria:

* Patients younger than 65 years old.
* Chronic kidney disease stages 1,2, and 3.
* Dialysis dependence
* History of kidney transplantation.
* Initial visit with the health care provider.
* Recent acute kidney injury.
* Patients who had been hospitalized for more than 2 months before the visit (because long hospitalization might affect the degree of frailty)
* Patients with myocardial infarction and cerebrovascular accident 3 months before the assessment
* Patients who are blind or with limb amputation.
* Patients who refuse to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults are diagnosed with advanced chronic kidney disease, namely, stage 4 and stage 5.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Time to death | 36 months
  The time from the assessment moment to death of an older adult with advanced CKD ( CKD stage 4 and 5).
Time to initiate dialysis. | 36 months
  The time from the assessment moment to start dialysis of an older adult with advanced CKD (

CONTACTS AND LOCATIONS:
Overall Officials: Hani Hussien, MD, Principal Investigator — University of Medicine and Pharmacy "Grigore T. Popa" - Iași
Locations (1):
- University of Medicine and Pharmacy "Grigore T. Popa", Iași, Romania